CLINICAL TRIAL: NCT02643420
Title: RAnDomized Trial of SPI-2012 Versus Pegfilgrastim in the Management of Chemotherapy Induced Neutropenia in Breast CANCEr Patients Receiving Docetaxel and Cyclophosphamide (TC) (ADVANCE)
Brief Title: SPI-2012 vs Pegfilgrastim in the Management of Neutropenia in Participants With Breast Cancer With Docetaxel and Cyclophosphamide (ADVANCE)
Acronym: ADVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-301
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Neutropenia; Breast Cancer
Keywords: Neutropenia; Breast Cancer; Long-acting Myeloid Growth Factor; Early Stage Breast Cancer; Docetaxel + Cyclophosphamide (TC) chemotherapy
MeSH Terms: conditions — Neutropenia; Breast Neoplasms | interventions — eflapegrastim; pegfilgrastim; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: SPI-2012 and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received SPI-2012 13.2 milligram (mg)/0.6 milliliter (mL) (3.6 mg Granulocyte Colony-Stimulating Factor [G-CSF]) fixed-dose subcutaneous (SC) injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy was administered on Day 1 of each cycle and included Docetaxel 75 mg/m^2 intravenous (IV) infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care.
  Interventions: Drug: SPI-2012; Drug: Docetaxel; Drug: Cyclophosphamide
- Arm 2: Pegfilgrastim and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received pegfilgrastim 6 mg SC injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy on Day 1 of each cycle included Docetaxel 75 mg/m^2 IV infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care.
  Interventions: Drug: Pegfilgrastim; Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: SPI-2012 — Single-use syringes for subcutaneous injection, administered on Day 2 of each cycle
  Other Names: Rolontis®; Eflapegrastim; (HM10460A)
  Arms: Arm 1: SPI-2012 and Docetaxel + Cyclophosphamide (TC)
Drug: Pegfilgrastim — Single-dose subcutaneous injection administered on Day 2 of each cycle
  Other Names: Neulasta®
  Arms: Arm 2: Pegfilgrastim and Docetaxel + Cyclophosphamide (TC)
Drug: Docetaxel — Standard therapy
  Other Names: Taxotere
Drug: Cyclophosphamide — Standard therapy
  Other Names: Cytoxan

SUMMARY:
The purpose of this study was to compare the efficacy of a single dose of SPI-2012 versus pegfilgrastim in participants with early-stage breast cancer receiving docetaxel and cyclophosphamide (TC), as measured by the duration of severe neutropenia (DSN) in Cycle 1.

DETAILED DESCRIPTION:
This was a Phase 3, randomized, open-label, active-controlled, multicenter study to compare the efficacy and safety of SPI-2012 vs pegfilgrastim in participants with breast cancer treated with TC chemotherapy.

Each cycle was 21 days. Four cycles were evaluated in this study. On Day 1 of each cycle, participants received TC chemotherapy. On Day 2 of each cycle, participants received study drug (SPI-2012 or pegfilgrastim).

ELIGIBILITY:
Key Inclusion Criteria:

* New diagnosis of histologically confirmed early-stage breast cancer (ESBC), defined as operable Stage I to Stage IIIA breast cancer
* Candidate for adjuvant or neoadjuvant TC chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
* Absolute neutrophil count (ANC) ≥ 1.5×10^9/L
* Platelet count ≥ 100×10^9/L
* Hemoglobin > 9 g/dL
* Creatinine clearance > 50 mL/min
* Total bilirubin ≤ 1.5 mg/dL
* Aspartate Aminotransferase per Serum Glutamic-Oxaloacetic Transaminase (AST/SGOT) and Alanine Aminotransferase per Serum Glutamic-Pyruvic Transaminase (ALT/SGPT) ≤ 2.5× Upper Limit of Normal (ULN).
* Alkaline phosphatase ≤ 2.0×ULN

Key Exclusion Criteria:

* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix) or life-threatening disease
* Locally recurrent or metastatic breast cancer
* Known sensitivity to E. coli -derived products or to any products to be administered during dosing
* Concurrent adjuvant cancer therapy
* Previous exposure to filgrastim, pegfilgrastim, or other G-CSF products in clinical development within 12 months prior to the administration of study drug
* Active infection, receiving anti-infectives, or any serious underlying medical condition that would impair ability to receive protocol treatment
* Prior bone marrow or stem cell transplant
* Use of any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study
* Radiation therapy within 30 days prior to enrollment
* Major surgery within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (81):
- United States (76):
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Arizona Clinical Research Center/ ACRC, Tucson, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NEA Baptist Clinic | Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Alta Bates Summit Medical Center, Berkeley, California
  - Precision Research Institute, LLC, Chula Vista, California
  - Compassionate Cancer Care Medical Group, Inc., Corona, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Pacific Shores Medical Group, Long Beach, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Emad Ibrahim, MD, Inc., Redlands, California
  - Compassionate Cancer Care Medical Group, Inc, Riverside, California
  - St Joseph Heritage Healthcare Institution, Santa Rosa, California
  - Wellness Oncology Hematology, West Hills, California
  - Oncology Institute of Hope and Innovation, Whittier, California
  - Omega Research Consultants LLC, DeBary, Florida
  - Pasco Pinellas Cancer Center, Holiday, Florida
  - AMPM Research Clinic, Miami, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Mid Florida Hematology and Oncology Centers, Orange City, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Bond Clinic, P.A., Winter Haven, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Dwight D. Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Clintell, Inc/Swedish Covenant Hospital, Chicago, Illinois
  - Joliet Oncology Hematology Associates, Joliet, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Swedish American Cancer Center, Rockford, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Floyd Memorial Cancer Center of Indiana, New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, Westville, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - West Ky Hematology & Oncology Group, PSC, Paducah, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Penobscot Bay Medical Center, Rockport, Maine
  - RCCA MD LLC/The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Reliant Medical Group, Worcester, Massachusetts
  - Quest Research Institute, Royal Oak, Michigan
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Freeman Health Systems, Joplin, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Southeast Nebraska Hematology & Oncology Consultants, PC, Lincoln, Nebraska
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - Mercy Health Youngstown LLC DBA, Youngstown, Ohio
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Associates in Hematology and Oncology, PC, Upland, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Bon Secours Saint Francis Cancer, Greenville, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - The West Clinic, PC, d/b/a West Cancer Center, Germantown, Tennessee
  - CHI St. Joseph Health Cancer Center, Bryan, Texas
  - Texas Oncology -Methodist Dallas Cancer Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology, PA, McAllen, Texas
  - Methodist Richardson Medical Center- Cancer Center, Richardson, Texas
  - Northern Utah Associates, Ogden, Utah
  - Delta Oncology Associates, Portsmouth, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (3):
  - CISSS de la Montérégie-Centre, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
- South Korea (2):
  - Cha Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Sinchon-dong, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 19 Jan 2016 to 31 Oct 2018. A total of 406 participants were randomized in the study.
Period: Overall Study
Arm/Group | Arm 1: SPI-2012 and Docetaxel + Cyclophosphamide (TC) | Arm 2: Pegfilgrastim and Docetaxel + Cyclophosphamide (TC)
Started | 196 | 210
Safety Population (Safety Population included all participants who had received at least one dose of any protocol specified drug (TC, SPI-2012, or pegfilgrastim).) | 197 (One participant was randomized to the Arm 2: Pegfilgrastim and TC but was inadvertently administered SPI-2012 on Cycle 1, Day 2 and was included in the Arm 1: SPI-2012 and TC for the Safety Population.) | 208
Completed | 142 | 145
Not Completed | 54 | 65
Not completed — Initiation of Non-Protocol Therapy for Breast Cancer | 6 | 12
Not completed — Withdrawal by Subject | 25 | 19
Not completed — Treatment with Additional Myeloid Growth Factors During Follow-up | 6 | 10
Not completed — Lost to Follow-up | 6 | 10
Not completed — Investigator Decision | 2 | 4
Not completed — Sponsor decision | 1 | 1
Not completed — Death | 0 | 2
Not completed — Reason not Specified | 8 | 7

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population included all participants who were randomized.
Groups:
- Arm 1: SPI-2012 and TC: Participants received SPI-2012 13.2 mg/0.6mL (3.6 mg G-CSF) fixed-dose SC injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy was administered on Day 1 of each cycle and included Docetaxel 75 mg/m^2 IV infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care.
- Arm 2: Pegfilgrastim and TC: Participants received pegfilgrastim 6 mg SC injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy on Day 1 of each cycle included Docetaxel 75 mg/m^2 IV infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care.
- Total: Total of all reporting groups
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC | Total
Number analyzed (Participants) | 196 | 210 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.12) | 59.0 (11.79) | 59.5 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 209 | 404
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 40 | 74
  Not Hispanic or Latino | 162 | 170 | 332
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 156 | 159 | 315
  Black or African American | 26 | 32 | 58
  Asian | 9 | 9 | 18
  American Indian or Alaska Native | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia (DSN) in Cycle 1
Description: DSN was defined as the number of days of severe neutropenia (absolute neutrophil count [ANC] <0.5×10^9/L), after the administration of study drug in Cycle 1.
Time Frame: Day 1 and Days 4-15 in Cycle 1 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
days | 0.20 (0.503) | 0.35 (0.683)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; Test type: Non-Inferiority — The margin of non-inferiority to be used in the study is 0.62 day. The non-inferiority of SPI-2012 to Pegfilgrastim was declared if the upper bound of 95% confidence interval (CI) of the difference in mean DSN between the treatment arms was <0.62 days; p < 0.0001, t-statistics; The p-values are based on the calculated t-statistics from the bootstrapped sample mean and standard deviation; Mean Difference (Final Values) = -0.148, 95% CI 2-sided [-0.266 to -0.031]

2. Secondary Outcome: Time to Absolute Neutrophil Count (ANC) Recovery in Cycle 1
Description: Time to ANC Recovery was defined as the time from chemotherapy administration until ANC increased to ≥1.5×10^9/L after the expected nadir within Cycle 1. Time to ANC recovery was assigned as 0 for participants whose ANC value never dropped below 1.5 x10^9/L.
Time Frame: Day 1 and Days 4, 15 in Cycle 1 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
days | 3.24 (3.565) | 3.49 (3.589)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; Test type: Superiority; p = 0.685, Negative binomial regression; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.43 to 0.94]

3. Secondary Outcome: Depth of Absolute Neutrophil Count (ANC) Nadir in Cycle 1
Description: Depth of ANC Nadir was defined as the lowest ANC value after administration of study drug (SPI-2012 or Pegfilgrastim) in Cycle 1.
Time Frame: Day 1 and Days 4, 15 in Cycle 1 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 191 | 196
10^9 ANC/L | 2.56 (3.086) | 2.53 (3.317)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; Test type: Superiority; p = 0.155, Asymptotic normality assumption; P-value was obtained based upon asymptotic normality assumption on the log10 transformed data; Median Difference (Final Values) = 1.2, 95% CI 2-sided [0.93 to 1.56]

4. Secondary Outcome: Number of Participants With Febrile Neutropenia (FN) in Cycle 1
Description: FN was defined as an oral temperature > 38.3 degrees Celsius (C) (101.0 degrees Fahrenheit [F]) or two consecutive readings of >=38.0 degrees C (100.4 degrees F) for 2 hours and ANC <1.0×10^9/L.
Time Frame: Day 1 and Days 4, 15 in Cycle 1 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
Participants | 4 | 2
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; Test type: Superiority; p = 0.435, Fisher Exact; Percent Difference = 1.1, 95% CI 2-sided [-8.6 to 10.8]

5. Secondary Outcome: Duration of Severe Neutropenia in Cycle 2, 3 and 4
Description: DSN was defined as the number of days of severe neutropenia (ANC <0.5×10^9 /L) from the first occurrence of an ANC below the threshold in Cycles 2, 3, and 4.
Time Frame: Days 1, 4, 7, 10, and 15 in cycles 2, 3, and 4 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
days
  Cycle 2 | 0.13 (0.383) | 0.09 (0.374)
  Cycle 3 | 0.11 (0.326) | 0.08 (0.273)
  Cycle 4 | 0.11 (0.362) | 0.09 (0.281)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; DSN in Cycle 2; Test type: Non-Inferiority — The margin of non-inferiority to be used in the study is 0.62 day. The non-inferiority of SPI-2012 to Pegfilgrastim was declared if the upper bound of 95% CI of the difference in mean DSN between the treatment arms was <0.62 days; p < 0.0001, t-statistics; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.032 to 0.116]
Statistical Analysis 2: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; DSN in Cycle 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, t-statistics; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.032 to 0.085]
Statistical Analysis 3: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; DSN in Cycle 4; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, t-statistics; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.036 to 0.089]

6. Secondary Outcome: Number of Participants With Neutropenic Complications in Cycle 1
Description: Neutropenic complications refer to hospitalizations due to neutropenic events and/or the use of anti-infectives due to neutropenia.
Time Frame: Day 1 and Days 4, 15 in Cycle 1 (each cycle was 21 days)
Population: The ITT population included all participants who was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
Participants | 8 | 8
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; Test type: Superiority; p = 1.000, Fisher Exact; Percent Difference = 0.3, 95% CI 2-sided [-9.5 to 10.0]

7. Secondary Outcome: Number of Participants With Febrile Neutropenia in Cycles 2, 3, and 4
Description: FN was defined as an oral temperature > 38.3 degrees C (101.0 degrees Fahrenheit [F]) or two consecutive readings of >=38.0 degrees C (100.4 degrees F) for 2 hours and ANC <1.0×10^9/L.
Time Frame: Days 1, 4, 7, 10, and 15 of Cycles 2, 3, and 4 (each cycle was 21 days)
Population: The ITT population included all participants who were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 196 | 210
Participants
  Cycle 2 | 1 | 1
  Cycle 3 | 4 | 1
  Cycle 4 | 2 | 0
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; FN in Cycle 2; Test type: Superiority; p = 1.000, Fisher Exact; Percent Difference = 0.0, 95% CI 2-sided [-9.7 to 9.8]
Statistical Analysis 2: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; FN in Cycle 3; Test type: Superiority; p = 0.201, Fisher Exact; Percent Difference = 1.6, 95% CI 2-sided [-8.2 to 11.3]
Statistical Analysis 3: Comparison: Arm 1: SPI-2012 and TC vs Arm 2: Pegfilgrastim and TC; FN in Cycle 4; Test type: Superiority; p = 0.232, Fisher Exact; Percent Difference = 1.0, 95% CI 2-sided [-8.7 to 10.8]

8. Secondary Outcome: Relative Dose Intensity (RDI) of TC (Docetaxel + Cyclophosphamide) in Cycles 1 to 4
Description: RDI was defined as the percentage of the planned dose that each participant actually received during the study, expressed as the total dose received, divided by the total dose planned and multiplied by 100. The planned dose was defined as the dose that would be given if no doses were missed and/or no dose reductions were made for the number of cycles started. The total planned dose was the sum of planned doses over all cycles.
Time Frame: Cycles 1 to 4 (each cycle was 21 days)
Population: Safety Population included all participants who received at least one dose of any protocol-specified drug (TC, SPI-2012 or pegfilgrastim). One participant was randomized to pegfilgrastim but was given SPI-2012 in Safety Population.
Measure: Mean (Standard Deviation); unit: percentage of planned dose
Arm/Group | Arm 1: SPI-2012 and TC | Arm 2: Pegfilgrastim and TC
Number analyzed (Participants) | 197 | 208
percentage of planned dose
  Docetaxel | 99.1 (5.47) | 98.1 (8.45)
  Cyclophosphamide | 99.3 (3.86) | 99.0 (4.33)

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product or study procedure, whether or not considered related to the medicinal product. A TEAE for Treatment Period is defined as adverse event with an onset date on or after the date of study drug administration through the end of treatment. TEAE for follow up is defined as any new onset or ongoing AE at the end of Treatment. SAE is defined as any AE which meets any of the following criteria: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in a persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, includes important medical events.
Time Frame: From the first dose of TC (Docetaxel + Cyclophosphamide) until 12 months after the last dose of study treatment (up to approximately 34 months)
Population: Safety Population included all participants who received at least one dose of any protocol-specified drug (TC, SPI-2012 or pegfilgrastim). One participant was randomized to pegfilgrastim but was given SPI-2012 in Safety Population. Data was summarized and reported separately for Treatment Period and Follow-up Period.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: SPI-2012 and TC -Treatment Period: Participants received SPI-2012 13.2 mg/0.6mL (3.6 mg G-CSF) fixed-dose SC injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy was administered on Day 1 of each cycle and included Docetaxel 75 mg/m^2 IV infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after the last study treatment or patient discontinuation.
- Arm 2: Pegfilgrastim and TC -Treatment Period: Participants received Pegfilgrastim 6 mg SC injection once per cycle on Day 2 of each cycle up to Cycle 4 (each cycle was 21 days), approximately 24-26 hours after TC chemotherapy administration. TC chemotherapy was administered on Day 1 of each cycle and included Docetaxel 75 mg/m^2 IV infusion and Cyclophosphamide 600 mg/m^2 IV infusion per institute's standard of care. All participants were followed for 35 (±5) days after the last study treatment or patient discontinuation.
- Arm 1: SPI-2012 and TC - Follow up Period; Arm 2: Pegfilgrastim and TC - Follow up Period: In addition to the treatment period, long-term safety follow-up continued for 12 months after last dose of study treatment.
Arm/Group | Arm 1: SPI-2012 and TC -Treatment Period | Arm 2: Pegfilgrastim and TC -Treatment Period | Arm 1: SPI-2012 and TC - Follow up Period | Arm 2: Pegfilgrastim and TC - Follow up Period
Number analyzed (Participants) | 197 | 208 | 197 | 208
Participants
  TEAE | 192 | 204 | 95 | 83
  SAE | 36 | 29 | 8 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of TC (Docetaxel + Cyclophosphamide) until 12 months after the last dose of study treatment (up to approximately 34 months)
Description: The safety population included all participants who had received at least one dose of any protocol specified drug (TC, SPI-2012, or pegfilgrastim). One participant was randomized to pegfilgrastim received SPI-2012 and was included in the Safety Population. Adverse events data was summarized and reported separately for the Treatment Period and Follow-up Period.
Arm/Group | Arm 1: SPI-2012 and TC -Treatment Period | Arm 2: Pegfilgrastim and TC -Treatment Period | Arm 1: SPI-2012 and TC - Follow up Period | Arm 2: Pegfilgrastim and TC - Follow up Period
All-Cause Mortality (participants affected / at risk) | 0/197 | 1/208 | 0/197 | 1/208
Serious Adverse Events (participants affected / at risk) | 36/197 | 29/208 | 8/197 | 2/208
Other Adverse Events (participants affected / at risk) | 192/197 | 203/208 | 92/197 | 82/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: SPI-2012 and TC -Treatment Period (N=197) | Arm 2: Pegfilgrastim and TC -Treatment Period (N=208) | Arm 1: SPI-2012 and TC - Follow up Period (N=197) | Arm 2: Pegfilgrastim and TC - Follow up Period (N=208)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 6 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Incision site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 0
Clostridium difficile sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 3 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Blood lactic acid increased (Investigations) | 1 | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: SPI-2012 and TC -Treatment Period (N=197) | Arm 2: Pegfilgrastim and TC -Treatment Period (N=208) | Arm 1: SPI-2012 and TC - Follow up Period (N=197) | Arm 2: Pegfilgrastim and TC - Follow up Period (N=208)
Fatigue (General disorders) | 120 | 124 | 14 | 8
Pyrexia (General disorders) | 45 | 45 | 0 | 1
Oedema peripheral (General disorders) | 36 | 28 | 3 | 3
Pain (General disorders) | 31 | 30 | 1 | 0
Asthenia (General disorders) | 16 | 18 | 1 | 0
Mucosal inflammation (General disorders) | 14 | 10 | 0 | 0
Chills (General disorders) | 11 | 9 | 1 | 0
Nausea (Gastrointestinal disorders) | 112 | 104 | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 87 | 86 | 3 | 3
Constipation (Gastrointestinal disorders) | 62 | 48 | 2 | 2
Vomiting (Gastrointestinal disorders) | 40 | 34 | 4 | 2
Stomatitis (Gastrointestinal disorders) | 26 | 25 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 20 | 25 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 20 | 17 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 11 | 15 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 13 | 12 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 13 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 71 | 70 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 36 | 20 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 40 | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 43 | 26 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 31 | 8 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 8 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 11 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 95 | 93 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 32 | 44 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 19 | 2 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 11 | 19 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 14 | 4 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 13 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 11 | 0 | 0
Lymphocyte count decreased (Investigations) | 80 | 74 | 2 | 0
White blood cell count decreased (Investigations) | 48 | 43 | 1 | 0
Neutrophil count decreased (Investigations) | 35 | 38 | 0 | 0
White blood cell count increased (Investigations) | 29 | 20 | 0 | 0
Platelet count decreased (Investigations) | 19 | 9 | 0 | 0
Neutrophil count increased (Investigations) | 13 | 11 | 0 | 0
Headache (Nervous system disorders) | 59 | 55 | 5 | 5
Dysgeusia (Nervous system disorders) | 36 | 29 | 0 | 0
Dizziness (Nervous system disorders) | 37 | 23 | 7 | 2
Neuropathy peripheral (Nervous system disorders) | 15 | 24 | 9 | 4
Neutropenia (Blood and lymphatic system disorders) | 67 | 65 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 51 | 39 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 19 | 22 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 13 | 14 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 5 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 26 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 31 | 7 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 25 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 0 | 3
Urinary tract infection (Infections and infestations) | 19 | 23 | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 38 | 31 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 22 | 21 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 13 | 0 | 1
Hot flush (Vascular disorders) | 21 | 22 | 15 | 16
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 4 | 10 | 7
Lacrimation increased (Eye disorders) | 9 | 9 | 0 | 0
Tachycardia (Cardiac disorders) | 11 | 10 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 10 | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02643420/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT02643420/SAP_001.pdf